CLINICAL TRIAL: NCT04687969
Title: Multimodal PET/MRI Machine Learning Approaches for Characterization of Solid Tumors
Brief Title: Multimodal Machine Learning Characterization of Solid Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Ciprian Catana, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ciprian Catana, MD, PhD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 20-048; R01CA218187 (NIH)
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Adenocarcinoma of Prostate; Radical Prostatectomy; Hepatocellular Carcinoma (HCC); Glioma; Renal Cell Carcinoma (RCC); Prostate Cancer
Keywords: Adenocarcinoma of Prostate; Radical Prostatectomy; Hepatocellular carcinoma (HCC); Glioma; Renal Cell Carcinoma (RCC); Prostate Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Glioma; Carcinoma, Renal Cell; Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- COHORT A: PROSTATE CANCER PATIENTS: Primary prostate cancer patients scheduled to undergo radical prostatectomy.
  * Twenty five (25) prostate cancer patients will undergo two [18F]DCFPyL PET/MRI scans and
  * Sixty (60) additional prostate cancer patients will undergo one [18F]DCFPyL PET/MRI scan.
  Interventions: Drug: [18F]DCFPyL; Radiation: PET/MRI scanner
- COHORT B: SOLID TUMOR PATIENTS: Patients with known or suspected solid tumors (hepatocellular carcinoma, glioma, clear cell renal carcinoma).
  Up to fifty (50) patients will undergo up to three [18F]DCFPyL PET/MRI scans
  Interventions: Drug: [18F]DCFPyL; Radiation: PET/MRI scanner

INTERVENTIONS:
Drug: [18F]DCFPyL — will either be administered by intravenous injection by bolus by a qualified nuclear medicine technician at the Martinos Center, or will be administered as part of a clinical PET/CT examination
  Other Names: positron emission tomography dye
Radiation: PET/MRI scanner — PET/MRI Scan with [18F]DCFPyL as directed by protocol
  Other Names: magnetic resonance imaging

SUMMARY:
This research study wants to develop advanced imaging methods to more accurately characterize prostate cancer or solid tumor aggressiveness.

This observational study involves [18F]DCFPyL positron emission tomography and magnetic resonance imaging (PET/MRI)

DETAILED DESCRIPTION:
This is an observational imaging study to evaluate the value of multimodal [18F]DCFPyL positron emission tomography and magnetic resonance imaging (PET/MRI) for solid tumor characterization and disease staging.

This research study involves:

* Screening visit, and 1-3 study Multimodal [18F]DCFPyL PET/MRI visits
* Two cohorts of participants will be enrolled in this study: primary prostate cancer patients and patients with known or suspected solid tumors (hepatocellular carcinoma, glioma, clear cell renal carcinoma)
* It is expected that about 135 people will take part in this research study

  * The PET dye used in this study is called [18F]DCFPyL. [18F]DCFPyL is approved by the U.S. Food and Drug administration (FDA).
  * The PET/MRI scanner was approved by the U.S. FDA.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:

  * Must have primary prostate cancer (e.g. adenocarcinoma of prostate) and deemed a candidate for radical prostatectomy as part of standard clinical care for Cohort A.
  * Must have evidence or be suspected of having HCC, Glioma and RCC for enrollment in Cohort B.
  * Age ≥18 years.

    --- Because no dosing or adverse event data are currently available on the use of [18F]DCFPyL in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
  * Participants must have adequate kidney function for gadolinium-based contrast administration as assessed by:

    * estimated or measured glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m2 for repeated administrations.
    * a single dose will be administered to subjects with a GFR between 30-60 mL/min/1.73 m2. Investigators will not repeat the gadolinium-based contrast agent administration until the renal function improves and the GFR is higher than 60 cc/min/1.73 m2. These subjects will not undergo examinations on consecutive days even if the renal function improves.
* Patient must be able to undergo MRI and PET scans.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the PET radiotracer, [18F]DCFPyL.
* Participants determined by the investigator(s) to be clinically unsuitable for the study.
* Patients who are not suitable to undergo MRI or PET or use gadolinium contrast due to:

  * Presence of ferromagnetic implants or implanted medical devices in body (i.e. cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body. tattoos near the eye, or steel implants)
  * Claustrophobia
  * Research-related radiation exposure exceeding current Massachusetts General Hospital (MGH) Radiology Department guidelines (i.e. 50 millisievert in the prior 12 months)
  * Inability to lie comfortably on bed inside the PET/MRI scanner
  * Body weight of > 300 lbs (weight limit of the MRI table)
  * Reduced renal function as determined by creatinine or GFR values defined above obtained within 30 days prior to registration
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must have primary prostate cancer (e.g. adenocarcinoma of prostate) and deemed a candidate for radical prostatectomy as part of standard clinical care for Cohort A.
  -- Must have evidence or be suspected of having HCC, Glioma and RCC for enrollment in Cohort B.
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of multimodal imaging in primary prostate cancer patients | 3 Days
  First tumor aggressiveness will be identified by binarizing the Gleason grade scores (GG ≥ 3+4). Binarized tumor aggressiveness obtained from the machine learning techniques will be then compared to the gold-standard, histopathology.

SECONDARY OUTCOMES:
Scan-rescan repeatability | 6 months
  Repeated measures analysis of covariance (ANCOVA) to evaluate statistical significance using a multilevel analysis to accommodate the nested structure of the data (longitudinal correlated data). Wilcoxon signed rank test will be used to assess for differences in each imaging parameter across visits. Spearman rank correlation will be used to test the correlation between [18F]-DCFPyL binding as measured by standardized uptake values (SUV) and Ktrans or SUV and cerebral blood flow (CBF). The false discovery rate will be used to adjust for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ciprian Catana, MD, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation